CLINICAL TRIAL: NCT06803524
Title: Antibody Persistence and Safety and Immunogenicity of a Second Booster Dose 10 Years After a First Booster Vaccination With a Single Dose Vaccination of aP Vaccine in Adults: A Phase IV, Open-label, Non-randomized, Follow-up Study
Brief Title: 10-year Follow-up After a Single Dose Acellular Pertussis Vaccination
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: BioNet-Asia Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor Emeritus, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TDA 202 10-year follow-up
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Pertussis
Keywords: TDA202; acellular pertussis vaccine; a second booster dose of Pertagen® as compared to Adacel®; antibody persistence at 10 years after vaccination; Pertagen; Boostagen; aP vaccine
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pertagen® vaccine (Experimental): Pertagen® vaccine, manufactured by BioNet-Asia Co., Ltd., Bangkok, Thailand. The vaccine is presented in pre-filled syringe, each containing one human dose (0.5 mL) of aP vaccine.
  Interventions: Biological: Pertagen® vaccine
- Adacel® vaccine (Experimental): Adacel® vaccine, manufactured by Sanofi Pasteur, Ltd, Toronto, Ontario, Canada. The vaccine is presented in a single-dose vial, each containing one human dose (0.5 mL) of Tdap vaccine.
  Interventions: Biological: Adacel® vaccine
- Boostagen® vaccine (Experimental): BIoNet Recombinant TdaP, each 0.5 mL dose of Boostagen (TdaP BioNet) contained 5 μg PTgen, 5 μg FHA, and 0.3 mg as aluminium cation.
  Interventions: Biological: Pertagen® vaccine

INTERVENTIONS:
Biological: Pertagen® vaccine — Pertagen® vaccine, manufactured by BioNet-Asia Co., Ltd., Bangkok, Thailand. The vaccine is presented in pre-filled syringe, each containing one human dose (0.5 mL) of aP vaccine.
  Arms: Boostagen® vaccine; Pertagen® vaccine
Biological: Adacel® vaccine — Adacel® vaccine, manufactured by Sanofi Pasteur, Ltd, Toronto, Ontario, Canada. The vaccine is presented in a single-dose vial, each containing one human dose (0.5 mL) of Tdap vaccine.
  Arms: Adacel® vaccine

SUMMARY:
This is a phase IV, open-label, non-randomized study to demonstrate superior immunogenicity and safety of a second booster dose of Pertagen® as compared to Adacel® at 10 years after the first booster vaccination and to evaluate the long-term persistence of specific antibodies induced by BioNet's recombinant aP (Pertagen®) and TdaP (Boostagen®) vaccines and a chemically-detoxified Tdap vaccine (Adacel®) at 10 years after the first booster in participants who were vaccinated in the phase II/III trial (Protocol No. TDA202).

DETAILED DESCRIPTION:
This is a phase IV, open-label, non-randomized study to demonstrate superior immunogenicity and safety of a second booster dose of Pertagen® as compared to Adacel® at 10 years after the first booster vaccination and to evaluate the long-term persistence of specific antibodies induced by BioNet's recombinant aP (Pertagen®) and TdaP (Boostagen®) vaccines and a chemically-detoxified Tdap vaccine (Adacel®) at 10 years after the first booster in participants who were vaccinated in the phase II/III trial (Protocol No. TDA202) conducted from July 2015 to November 2016. Only those who were enrolled in the initial TDA202 study and had completed TDA202 1-year follow-up will be recruited for this 10-year follow-up study.

Participants from all 3 vaccine groups (i.e., participants who had received a single dose of one of the 3 study vaccines (Boostagen®, Pertagen®, or Adacel®) and completed 1-year follow-up visit at Day 336±28 days during the TDA202 study will be called in for informed consent process at Visit 0 (Screening) at approximately 10 years (range, 9.5-10 years) following vaccination.

At Visit 0, Screening visit, participants who have signed the written Informed Consent Forms will be screened for general health status (medical history, medication history, immunization history, history of receiving blood, blood component, immunoglobulin, immunosuppressive drugs or systemic corticosteroid, vital signs and physical examination) and those who fulfill the pre-defined inclusion criteria without meeting any exclusion criteria will be enrolled into the study. The screening visit and Visit 1 (Day 0) can be completed on the same day. Once enrolled, a blood sample (approx. 5 mL) will be taken from all participants at Visit 1 (before second booster vaccination) and at Visit 2 (28 days after second booster vaccination) as shown in the diagram below (Figure 1).

At Visit 1, Day 0 (enrollment and second booster vaccination), a blood sample (approx. 5 mL) will be taken from all enrolled participants. After blood collection, the participants who received Pertagen® and Boostagen® in the initial TDA202 study will be administered a single intramuscular injection of a second booster dose of Pertagen®. The participants who have received Adacel® in the initial TDA202 study will be given a single intramuscular injection of a second booster dose of Adacel® (Table 1). Composition of booster vaccines are presented in Table 2. The vaccine preparation and administration will be performed by appropriately trained study team and study nurses, respectively, who are delegated by the Principal Investigator.

If a participant does not complete screening visit and Visit 1 (Day 0) on the same day, the screening process for general health status (medical history, medication history, immunization history, history of receiving blood, blood component, immunoglobulin, immunosuppressive drugs or systemic corticosteroid, vital signs and physical examination), urine pregnancy test for female participants with childbearing potential and inclusion and exclusion criteria will be assessed again at Visit 1.

Brief description of the study design for TDA202 10-year follow-up study:

This is a phase IV, open-label, non-randomized study to demonstrate superior immunogenicity and safety of a second booster dose of Pertagen® as compared to Adacel® at 10 years after the first booster vaccination and to evaluate the long-term persistence of specific antibodies induced by BioNet's recombinant aP (Pertagen®) and TdaP (Boostagen®) vaccines and a chemically-detoxified Tdap vaccine (Adacel®) at 10 years after the first booster in participants who were vaccinated in the phase II/III trial (Protocol No. TDA202) conducted from July 2015 to November 2016. Only those who were enrolled in the initial TDA202 study and had completed TDA202 1-year follow-up will be recruited for this 10-year follow-up study.

Participants from all 3 vaccine groups (i.e., participants who had received a single dose of one of the 3 study vaccines (Boostagen®, Pertagen®, or Adacel®) and completed 1-year follow-up visit at Day 336±28 days during the TDA202 study will be called in for informed consent process at Visit 0 (Screening) at approximately 10 years (range, 9.5-10 years) following vaccination.

At Visit 0, Screening visit, participants who have signed the written Informed Consent Forms will be screened for general health status (medical history, medication history, immunization history, history of receiving blood, blood component, immunoglobulin, immunosuppressive drugs or systemic corticosteroid, vital signs and physical examination) and those who fulfill the pre-defined inclusion criteria without meeting any exclusion criteria will be enrolled into the study. The screening visit and Visit 1 (Day 0) can be completed on the same day. Once enrolled, a blood sample (approx. 5 mL) will be taken from all participants at Visit 1 (before second booster vaccination) and at Visit 2 (28 days after second booster vaccination) as shown in the diagram below (Figure 1).

At Visit 1, Day 0 (enrollment and second booster vaccination), a blood sample (approx. 5 mL) will be taken from all enrolled participants. After blood collection, the participants who received Pertagen® and Boostagen® in the initial TDA202 study will be administered a single intramuscular injection of a second booster dose of Pertagen®. The participants who have received Adacel® in the initial TDA202 study will be given a single intramuscular injection of a second booster dose of Adacel® (Table 1). Composition of booster vaccines are presented in Table 2. The vaccine preparation and administration will be performed by appropriately trained study team and study nurses, respectively, who are delegated by the Principal Investigator.

If a participant does not complete screening visit and Visit 1 (Day 0) on the same day, the screening process for general health status (medical history, medication history, immunization history, history of receiving blood, blood component, immunoglobulin, immunosuppressive drugs or systemic corticosteroid, vital signs and physical examination), urine pregnancy test for female participants with childbearing potential and inclusion and exclusion criteria will be assessed again at Visit 1.

Table 1: Vaccine groups and booster dose vaccination Vaccine group in Initial TDA202 study Second booster vaccination at Day 0 Total number of participants (N) per vaccine group Pertagen® and Boostagen® Pertagen® 84 Adacel® Adacel® 42 After the second booster vaccination, participants will be observed at the study site for at least 30 minutes to monitor for any immediate post-immunization reactions. Safety and reactogenicity in the participants will be assessed until end of study. The diary cards will be distributed to the participants to record post-immunization solicited local and systemic adverse events (AEs) until Day 7 and unsolicited AEs, serious adverse events (SAEs), and concomitant medications until Day 28 following vaccination. The study staff will contact the participants by phone on Day 7 (+4 days) to enquire on health status and to remind them to record any solicited local and systemic AEs, unsolicited AE, SAE and concomitant medications in the diary card.

At Visit 2, Day 28 (+7 days), participants will return to the study site for blood sample collection (approx. 5 mL), reconciliation of information in the diary card, and any reported AEs, SAEs and concomitant medications.

Safety and reactogenicity will be assessed until end of study. Solicited local and systemic AEs will be collected until Day 7 after the second booster vaccination. Unsolicited Adverse Events (AEs) and Serious Adverse Events (SAEs) will be collected until Visit 2 (Day 28) after the second booster vaccination. Visit 2 is considered the end of study.

Blood samples collected from all participants at Day 0 (Visit 1) and Day 28 (Visit 2) will be processed for serum preparation. Serum samples will be stored at the laboratory at the study site and will be further shipped to BioNet-Asia Human Serology Laboratory where immunogenicity testing will be performed. At Day 0 (Visit 1) and Day 28 (Visit 2), ELISA testing to detect antibodies against pertussis toxoid (PT), filamentous hemagglutinin (FHA) and PT neutralizing assay in Chinese Hamster Ovary (CHO) cells will be performed for all enrolled participants. At Day 0 (Visit 1), ELISA testing to detect antibodies against tetanus toxoid (TT) and diphtheria toxoid (DT) will be performed for participants who received Boostagen® and Adacel® in TDA202 initial study.

Data management and statistical analysis will be performed by the Center of Excellence for Biomedical and Public Health Informatics (BIOPHICS), Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for inclusion if ALL of the following apply at the time of screening:

1. Having participated in the initial TDA202 study, received a single dose of one of the 3 study vaccines, and completed 1-year follow-up visit;
2. Written informed consent is obtained prior to study entry;
3. Healthy, as established by pertinent medical history and physical examination;
4. Capable of complying with study procedures and willing to provide with a blood sample;
5. For women with childbearing potential (i.e., urine pregnancy test will not be performed in females who have undergone sterilisation, hysterectomy or who are post-menopausal), must have a negative urine pregnancy test at enrollment and willing to take reliable birth control measures for one month following vaccination.

Exclusion Criteria:

A participant with following criteria at screening will not be eligible for participation:

1. Having received any pertussis vaccine since completion of 1-year follow-up visit in the initial TDA202 study;
2. Having experienced physician-diagnosed pertussis since completion of 1-year follow-up visit in the initial TDA202 study prior to enrollment;
3. Pregnant or breast-feeding women or female participants who intend to become pregnant during study period;
4. History of any significant medical illness such as, but not limited to, immune deficiency, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic, renal, or endocrine disorder, splenic or thymic functional abnormality as determined by the investigator based on medical history and physical examination that may interfere with the participant's safety and evaluation of investigational vaccines in this study;
5. History of allergy or hypersensitivity to any vaccine (including its component);
6. History of any serious adverse event or neurological adverse event after vaccination;
7. History of receiving blood or blood component or immunoglobulin within 3 months prior to enrollment;
8. History of receiving immunosuppressive drugs or systemic corticosteroid (>0.5 mg/kg of prednisolone or equivalent for more than 14 days) within 3 months prior to enrollment;
9. Having received any other vaccines within 28 days prior to enrollment (3 months for live- attenuated vaccines);
10. Plan to receive any other vaccine or plan to participate in another clinical trial with intervention during the study period;
11. A known bleeding diathesis or any condition that may be associated with a prolonged bleeding time resulting in a problem with intramuscular injection;
12. Any progressive or severe neurological disorder such as seizure disorder or Guillain-Barré syndrome;
13. History of any illness or clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the volunteers due to participation in the study
14. Fever as defined by body temperature ≥ 38°C at the time of enrollment (This is a temporary exclusion criterion).

Remark: If fever occurs at screening visit, the participant may be rescreened and enrolled at a later date at the discretion of the investigator, or withdrawn at the discretion of the investigator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To demonstrate superiority at 28 days post-booster vaccination with one dose of Pertagen® as compared to Adacel®. | Day 28
  Geometric mean concentration (GMC) of anti-PT and anti-FHA antibodies measured at baseline (before second booster vaccination) and 28 days following vaccination.

SECONDARY OUTCOMES:
Immunogenicity endpoints at 28 days post-booster vaccination with one dose of Pertagen® as compared to Adacel®. | Day 28
  • GMC of PT neutralizing antibody (PTNA) measured at baseline (before second booster vaccination) and 28 days following vaccination.
Immunogenicity endpoints at 28 days post-booster vaccination with one dose of Pertagen® as compared to Adacel®. | Day 28
  • Seroconversion rates as defined by proportion of participants with antibody concentrations ≥ 4-fold increase with respect to baseline (before first and second booster vaccination) of anti-PT and anti-FHA, and PT- neutralizing antibodies at 28 days after booster dose vaccination.
Immunogenicity endpoints at 28 days post-booster vaccination with one dose of Pertagen® as compared to Adacel®. | Day 28
  • Seropositive rates as defined by proportion of participants with antibody concentrations > 5 IU/mL for anti-PT and anti-FHA, and PT-neutralizing antibodies at baseline (before first and second booster vaccination) and 28 days after booster dose vaccination.
Immunogenicity endpoints at 28 days post-booster vaccination with one dose of Pertagen® as compared to Adacel®. | Day 28
  • Booster response rates as defined by proportion of participants with antibody concentrations >20 IU/mL for anti-PT and anti-FHA, and PT-neutralizing antibodies at baseline (before first and second booster vaccination) and 28 days after booster dose vaccination.
Immunogenicity endpoints at 28 days post-booster vaccination with one dose of Pertagen® as compared to Adacel®. | Day 28
  • The proportion of participants with cut-off levels of anti-PT, anti-FHA and PT-neutralizing antibodies (i.e, ≥ 5, > 5, ≥ 10, ≥ 20, ≥ 30, ≥ 40, ≥ 50, ≥ 80, ≥ 100, ≥ 120 IU/mL) in Pertagen® and Adacel® at baseline (before first and second booster vaccination) and 28 days after booster dose vaccination.
Immunogenicity endpoints for antibody response before second booster vaccination at 10 years after a single dose vaccination of Boostagen® and Pertagen® as compared to Adacel® from initial TDA202 study | 10 years safter vaccination
  • GMCs of anti-PT, anti-FHA and PT-neutralizing antibodies in all vaccine groups and GMCs of anti-TT and anti-DT antibodies in Boostagen® and Adacel® at 10 years after vaccination
Immunogenicity endpoints for antibody response before second booster vaccination at 10 years after a single dose vaccination of Boostagen® and Pertagen® as compared to Adacel® from initial TDA202 study | 10 years safter vaccination
  • Seropositive rates as defined by proportion of participants with antibody concentrations >5 IU/mL for anti-PT and anti-FHA, and PT-neutralizing antibodies at 10 years after vaccination
Immunogenicity endpoints for antibody response before second booster vaccination at 10 years after a single dose vaccination of Boostagen® and Pertagen® as compared to Adacel® from initial TDA202 study | 10 years safter vaccination
  • Booster response rates as defined by proportion of participants with antibody concentrations >20 IU/mL for anti-PT and anti-FHA, and PT neutralizing antibodies at 10 years after vaccination
Immunogenicity endpoints for antibody response before second booster vaccination at 10 years after a single dose vaccination of Boostagen® and Pertagen® as compared to Adacel® from initial TDA202 study | 10 years safter vaccination
  • Seroconversion rates as defined by proportion of participants with antibody concentrations ≥ 2-fold increase with respect to baseline of anti-PT and anti-FHA, and PT-neutralizing antibodies at 10 years after vaccination
Immunogenicity endpoints for antibody response before second booster vaccination at 10 years after a single dose vaccination of Boostagen® and Pertagen® as compared to Adacel® from initial TDA202 study | 10 years safter vaccination
  • Seroconversion rates as defined by proportion of participants with antibody concentrations ≥ 4-fold increase with respect to baseline, of anti-PT and anti-FHA, and PT-neutralizing antibodies at 10 years after vaccination
Immunogenicity endpoints for antibody response before second booster vaccination at 10 years after a single dose vaccination of Boostagen® and Pertagen® as compared to Adacel® from initial TDA202 study | 10 years safter vaccination
  • Seroprotection rate as defined by proportion of participants with antibody concentrations > 0.1 IU/mL of anti-TT and anti-DT antibodies in Boostagen® and Adacel® vaccine groups at 10 years after vaccination. The proportion of participants with cut-off levels of anti-PT, anti-FHA and PT-neutralizing antibodies (i.e, ≥ 5, > 5, ≥ 10, ≥ 20, ≥ 30, ≥ 40, ≥ 50, ≥ 80, ≥ 100, ≥ 120 IU/mL) in Pertagen®, Boostagen® and Adacel® at 10 years after vaccination
Safety endpoints at 28 days post-booster vaccination with one dose of Pertagen® and Adacel® | From Day 0 to Day 7
  • Percentage of participants with solicited local and systemic AEs reported within 7 days after booster vaccination
Safety endpoints at 28 days post-booster vaccination with one dose of Pertagen® and Adacel® | From Day 0 to Day 28
  • Percentage of participants with unsolicited AEs reported from the day of booster vaccination through 28 days following booster vaccination
Safety endpoints at 28 days post-booster vaccination with one dose of Pertagen® and Adacel® | From Day 0 to Day 28
  • Percentage of participants with SAEs reported from the day of booster vaccination through 28 days following booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Principal Investigator — Vaccine trial Centre
Locations (2):
- Thailand (2):
  - Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok Metropolis
  - Vaccine Trial Centre, Ratchathewi, Bangkok Metropolis

IPD SHARING:
Plan to Share IPD: No